CLINICAL TRIAL: NCT01335152
Title: Coping With Breast Cancer and Treatment: An E-Learning Course for Skills and Strategies
Brief Title: Online Stress Management and Coping Skills Training for Women With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Talaria, Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA106154; 5R44CA106154-03 (NIH)
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: stress; depression; anxiety; web; internet; coping
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders | interventions — Coping Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Web-based workbook (Experimental): Participants will use one chapter of the web-based workbook each week for 10 weeks. The workbook consists of stress management education, cognitive behavioral interventions and relaxation training exercises.
  Interventions: Behavioral: Coping with Breast Cancer web-based workbook
- Waitlist control group (No Intervention): Participants will no intervention for the first 10 weeks of the study and then will receive the web-based intervention.

INTERVENTIONS:
Behavioral: Coping with Breast Cancer web-based workbook — 10 chapter web-based workbook that teaches stress management, cognitive behavioral coping skills and relaxation training.
  Other Names: Stress management; Coping with Cancer; Cancer Coping; Online workbook
  Arms: Web-based workbook

SUMMARY:
Stress Management interventions have been shown to decrease cancer-related distress, foster emotional growth and improve immune functioning during treatment for breast cancer.

This study will evaluate an online version of a stress management intervention for women with early stage breast cancer. Each chapter of the 10-week intervention include self-assessment and targeted feedback, education, interactive learning exercises -- all tailored to the needs of women with early stage breast cancer. In addition, guided writing exercises will promote emotional expression and a discussion board will encourage group support.

The web-based intervention is being evaluated in a randomized clinical trial with a sample of 120 women with early stage breast cancer. Women will be randomly assigned to use the 10-week intervention with biweekly telephone assessments or to the telephone assessments alone.

DETAILED DESCRIPTION:
Stress Management interventions have been shown to decrease cancer-related distress, foster emotional growth and improve immune functioning during treatment for breast cancer.

This study will evaluate an online version of a stress management intervention for women with early stage breast cancer. Each chapter of the 10-week intervention include self-assessment and targeted feedback, education, interactive learning exercises -- all tailored to the needs of women with early stage breast cancer. In addition, guided writing exercises will promote emotional expression and a discussion board will encourage group support.

The web-based intervention is being evaluated in a randomized clinical trial with a sample of 120 women with early stage breast cancer. Women will be randomly assigned to use the 10-week intervention with biweekly telephone assessments or to the telephone assessments alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage 0, I, II or III breast cancer within past 18 months
* Elevated stress, distress or negative mood
* Access at least 1.5 - 2 hours per week to a computer with audio capabilities that is connected to the internet
* Ability to read, write, and speak English at a sixth grade level
* Access to a telephone and an active e-mail account

Exclusion Criteria:

* Cancer diagnosis is a recurrence
* Diagnosis of schizophrenia
* Use of anti-psychotic medication
* Diagnosis of bipolar disorder without use of mood stabilizing medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
PHQ GAD-7 - Anxiety | baseline, post-intervention, follow-up
  7-item self-report questionnaire measureing anxiety.
CES-D 10 | baseline, post-intervention, follow-up
  10 item self-report measure of depression.
FACT-B: Functional Assessment of Cancer Therapy - Breast | baseline, post-intervention, follow-up
  44 item self-report measure of health related quality of life for breast cancer patients.

SECONDARY OUTCOMES:
Revised Impact of Event Scale | baseline, post-intervention, follow-up
  22 item self-report measure of intrusive thoughts and avoidance of cancer-related thoughts.
Benefit Finding Scale for breast cancer | baseline, post-intervention, follow-up
  17-item self-report measure of finding positive impact of negative events.
CANCER BEHAVIOR INVENTORY (CBI-B) | baseline, post-intervention, follow-up
  16-item self-report measure of self-efficacy for coping with cancer and cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly M Carpenter, PhD, Principal Investigator — Talaria, Inc
Locations (1):
- Talaria, Inc, Seattle, Washington, United States